CLINICAL TRIAL: NCT05477485
Title: Antiretroviral Improvement Among Medicaid Enrollees (AIMS): An Insurance-based Data to Care Initiative for Medicaid Enrollees in Virginia
Brief Title: Antiretroviral Improvement Among Medicaid Enrollees
Acronym: AIMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient rate of accrual
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH); Virginia Department of Medical Assistance Services - Virginia Medicaid (Unknown); Virginia Department of Health (Other Government); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20018229; U01PS005192 (NIH)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other): Usual Care participants will receive standard state-level care for missing ART prescription refill(s) for Virginia Medicaid enrollees with HIV.
  Interventions: Other: No Intervention/Usual care
- AIMS program - patient (Experimental): Participants will receive patient-level support. Support will come from the participant's provider, pharmacy, managed-care organization or the community.
  Interventions: Behavioral: Experimental: AIMS program - patient

INTERVENTIONS:
Behavioral: Experimental: AIMS program - patient — Patient-level support will be offered to eligible Virginia Medicaid enrollees who have a late ART prescription refill(s) by >30 days. Support will come from the provider, pharmacy, managed care organization or the community. Patient-level support will involve direct linkages and referrals for participants with a late ART prescription refill(s) >30-60 days. Support will intensify as the gap in ART prescription(s) fills increases. For those with a late ART prescription refill(s) for >60 days, added patient-level support will include warm health technology via PositiveLinks, a mobile app program promoting better health through self-monitoring tools, educational resources, direct messaging with program staff and a confidential user community board.
  Arms: AIMS program - patient
Other: No Intervention/Usual care — Participants in the usual care arm will receive standard state-level care for late ART prescription refill(s) for Virginia Medicaid enrollees living with HIV.
  Arms: Usual Care

SUMMARY:
This study will evaluate whether a new program will affect how often human immunodeficiency virus (HIV) antiretroviral therapy (ART) prescriptions are filled and whether the program improves the health of people living with HIV.

DETAILED DESCRIPTION:
Virginia Commonwealth University and study collaborators are working together to learn about challenges that Virginia Medicaid members have in taking their prescribed medication. To do this, the researchers are implementing and evaluating a program called Antiretroviral Improvement among Medicaid enrolleeS (AIMS). This program is designed to support members to fill ART prescriptions.

The program involves supporting Medicaid members with HIV directly by talking to them about challenges with filling their ART prescriptions and linking them to resources that can help with those challenges. Some members will be offered access to warm health technology support.

The researchers think this support may increase how often ART prescriptions are filled and hope that the AIMS program can improve individuals' health and increase HIV viral suppression.

ELIGIBILITY:
Inclusion criteria:

* Current enrollment in Virginia Medicaid;
* Continuous Virginia Medicaid enrollment for the preceding 9 or more months;
* Current age 19-64 years;
* Identified as living with HIV according to an HIV case identification algorithm;
* Non-dual eligible for Medicare;
* History of ART prescription claim(s) within the past 12 months;
* Prior ART prescription claim, with claims for the most recent ART prescription refill(s) >30 days late.

Exclusion criteria:

* Record of non-Medicaid health insurance or other health care service payer in past 3 months;
* New prescription claim(s) within 30 days for within-class ART drug(s) not previously prescribed;
* Service claim(s) for resistance testing and other ART prescription claim(s) within 30 days of most recent late ART prescription(s) for ART drug(s) not previously prescribed;
* Enrollee's linked HIV provider practices at a healthcare facility offering PositiveLinks;
* No record in the Virginia HIV surveillance data;
* Non-English speaking.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April D Kimmel, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimmel AD, Byrd KK, Stirratt M, Harris D, Stallings R, Bono RS, Mitchell A, Dillingham R, Palmer C, Popoff E, Pan Z, Ingersoll K, Dahman B; AIMS study team. Study Protocol(s) for Antiretroviral Improvement among Medicaid EnrolleeS (AIMS): A Cluster-Randomized Controlled Trial Leveraging Real-time Administrative Claims to Support Antiretroviral Prescription Adherence. Contemp Clin Trials. 2025 Jul;154:107959. doi: 10.1016/j.cct.2025.107959. Epub 2025 May 18. PMID 40393614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the intervention (AIMS program-patient arm) occurred April 2023-May 2024, with n=4 enrolled in the intervention. Recruitment for the Usual Care arm does not apply. The study design was such that the Usual Care arm would be constructed after follow-up on the intervention. As the trial was terminated due to insufficient rate of accrual for the intervention, no such sample was constructed. No data were collected for the Usual Care arm (n=0); there are no data to analyze or report.
Groups:
- Usual Care: Usual Care participants will receive standard state-level care for missing ART prescription refill(s) for Virginia Medicaid enrollees with HIV.
  No Intervention/Usual care: Participants in the usual care arm will receive standard state-level care for late ART prescription refill(s) for Virginia Medicaid enrollees living with HIV. Recruitment for the Usual Care group does not apply. The Usual Care group was a comparison group to be constructed from existing data. The trial ended with an insufficient rate of accrual for the AIMS program-patient (intervention) group, no sample was constructed. No data was collected for the usual care arm (n=0), there is no data to report.
Period: Overall Study
Arm/Group | Usual Care | AIMS program - patient
Started | 0 | 4
Completed | 0 | 0
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Usual Care group was not constructed because the trial was terminated. The study design was such that the Usual Care arm would be constructed after follow-up on the intervention (AIMS program - patient arm). No data were collected for the Usual Care arm (n=0); there are no data to analyze or report.
Groups:
- Usual Care: No Intervention/Usual care: Participants in the usual care arm will receive standard state-level care for late ART prescription refill(s) for Virginia Medicaid enrollees living with HIV. Recruitment for the Usual Care group does not apply. The Usual Care group was a comparison group to be constructed from existing data. The trial ended with an insufficient rate of accrual for the AIMS program-patient (intervention) group, no sample was constructed. No data was collected for the usual care arm (n=0), there is no data to report.
- Total: Total of all reporting groups
Arm/Group | Usual Care | AIMS program - patient | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 45 (10.6) | 45 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2
  Male |  | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 4 | 4
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 2 | 2
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Virally Suppressed
Description: HIV viral load data come from Virginia Department of Health (VDH) routine surveillance. Viral load data indicate whether or not an individual was virally suppressed, i.e., the level of HIV in a blood sample was less than the detectable limit.
Time Frame: 3 months
Population: Data for this outcome measure would have been obtained through data reports made available through the Virginia Department of Health (VDH). At the time of this outcome measure, when data would have been collected, there were no reports from VDH. Therefore, no primary outcome data were available to be collected for all enrolled participants in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | AIMS program - patient
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

2. Secondary Outcome: Number and Percentage of Participants Reinitiating Late Antiretroviral Therapy (ART) Prescription
Description: Data source is prescription claim(s) for antiretroviral therapy (ART) prescription(s) made available through Virginia Medicaid. Participants will be considered as reinitiating if they have a filled ART prescription after study enrollment.
Time Frame: 3 months
Population: 4 subjects enrolled in the intervention (AIMS program - pt arm, n=4). No participants were enrolled into the usual care arm, and therefore, no data were collected for this outcome measure for that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | AIMS program - patient
Number analyzed (Participants) | 0 | 4
Participants | 0 | 4

3. Secondary Outcome: Antiretroviral Therapy (ART) Adherence
Description: Data source is prescription claim(s) for antiretroviral therapy (ART) made available through Virginia Medicaid. Participants will be considered adherent if their ART prescription claim(s) cover >90% of enrolled coverage days.
Time Frame: 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | AIMS program - patient
Number analyzed (Participants) | 0 | 4
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Description: Medical adverse events do not apply.
  Adverse events consist of emotional or psychological distress during the AIMS program-patient intervention phone call or during use of the optional PositiveLinks app.
  Adverse events do not apply to the Usual Care group.
Arm/Group | Usual Care | AIMS program - patient
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4

LIMITATIONS AND CAVEATS:
Four participants enrolled in the intervention (AIMS program - patient arm, n=4). For the primary outcome, all enrolled participants were lost to follow-up. Primary outcome data were not available. No participants were enrolled in the usual care arm (n=0), and therefore, no data were collected for the outcome measures for that arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05477485/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05477485/ICF_002.pdf